CLINICAL TRIAL: NCT01247935
Title: Electroacupuncture and Trancutaneous Electrical Nervous Stimulation Analgesia for Colonoscopy: a Prospective, Randomized, Controlled Study
Brief Title: Electroacupuncture and Trancutaneous Electrical Nervous Stimulation (TENS) for Colonoscopy Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Per I Servizi Sanitari N. 2 Isontina (Other)
Responsible Party: Corrado Thomann, Azienda per i Servizi Sanitari n. 2 Isontina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 34115/14
Record Dates: First submitted 2010-11-12; First posted 2010-11-25 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2010-06

CONDITIONS: Pain
Keywords: Pain; Acupuncture; Transcutaneous electrical nerve stimulation; Colonoscopy
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy; Electroacupuncture; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture (Experimental): Electrostimulation at 5 Hz in GI4, ST36, MP6, MP9 starting 20 minutes before colonoscopy
  Interventions: Other: Acupuncture
- transcutaneous electrical stimulation (Experimental): Electrostimulation at 5 Hz in GI4, ST36, MP6, MP9 starting 20 minutes before colonoscopy
  Interventions: Other: Transcutaneous electrical stimulation
- Control (No Intervention): patient are monitored for pain and discomfort
  Interventions: Other: Control

INTERVENTIONS:
Other: Acupuncture — Electrostimulation at 5 Hz in GI4, ST36, MP6, MP9 starting 20 minutes before colonoscopy
  Other Names: Electroacupuncture
  Arms: Acupuncture
Other: Transcutaneous electrical stimulation — Electrostimulation at 5 Hz in GI4, ST36, MP6, MP9 starting 20 minutes before colonoscopy
  Other Names: TENS
  Arms: transcutaneous electrical stimulation
Other: Control — Patients are monitored for pain and discomfort
  Other Names: No treatment (only sedative drugs if request)
  Arms: Control

SUMMARY:
To compare the effectiveness of acupuncture and transcutaneous electrical nervous stimulation (TENS) in reducing patient's discomfort during colonoscopy

DETAILED DESCRIPTION:
Evaluation patient's pain and discomfort during colonoscopy, using two non invasive analgesic methods.

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for colonoscopy and in whom deep sedation was not planned will be included in the study

Exclusion Criteria:

* age > 80 and less than 18 years old, severe cardiac or pulmonary disease, anticoagulant, benzodiazepines, antidepressants, opiates therapies, severe cognitive impairment, uncontrolled hypertension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of patients' discomfort and pain during and at the end of colonoscopy both in acupuncture group and in TENS group compare with controls. | During colonoscopy, we'll evaluate pain at colorectal, left, trasversal and right colon position of colonscope. At the end of colonoscopy, before discharge, we' ll evaluate patient's general discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Thomann, MD, Principal Investigator — ICU Gorizia Hospital
Locations (1):
- Presidio Ospedaliero di Gorizia, Gorizia, Italy

REFERENCES:
- [Background] Sung JJ. Acupuncture for gastrointestinal disorders: myth or magic. Gut. 2002 Nov;51(5):617-9. doi: 10.1136/gut.51.5.617. PMID 12377792
- [Background] Camilleri M. Editorial: is adequate relief fatally flawed or adequate as an end point in irritable bowel syndrome? Am J Gastroenterol. 2009 Apr;104(4):920-2. doi: 10.1038/ajg.2009.20. Epub 2009 Mar 17. PMID 19293789
- [Background] Han JS. Acupuncture and endorphins. Neurosci Lett. 2004 May 6;361(1-3):258-61. doi: 10.1016/j.neulet.2003.12.019. PMID 15135942
- [Background] Fanti L, Gemma M, Passaretti S, Guslandi M, Testoni PA, Casati A, Torri G. Electroacupuncture analgesia for colonoscopy. a prospective, randomized, placebo-controlled study. Am J Gastroenterol. 2003 Feb;98(2):312-6. doi: 10.1111/j.1572-0241.2003.07231.x. PMID 12591047
- [Background] Robinson R, Darlow S, Wright SJ, Watters C, Carr I, Gadsby G, Mayberry J. Is transcutaneous electrical nerve stimulation an effective analgesia during colonoscopy? Postgrad Med J. 2001 Jul;77(909):445-6. doi: 10.1136/pmj.77.909.445. PMID 11423594